CLINICAL TRIAL: NCT05644951
Title: A Prospective, Multi-center, Single-arm Study for Unresectable Malignant Gastric Outlet Obstruction With EUS-guided Double-balloon-occluded Gastrojejunostomy Bypass
Brief Title: Clinical Trial of EPASS With Hot AXIOS System
Acronym: PASSAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E7127
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hot AXIOS system (Experimental): Hot AXIOS system (20 mm diameter stent)
  Interventions: Device: Hot AXIOS system used for EPASS

INTERVENTIONS:
Device: Hot AXIOS system used for EPASS — EUS-guided double-balloon-occluded gastrojejunostomy bypass with Hot AXIOS system

SUMMARY:
A prospective, multi-center, single-arm study for unresectable malignant gastric outlet obstruction with EUS-guided double-balloon-occluded gastrojejunostomy bypass (EPASS)

DETAILED DESCRIPTION:
Primary objective is to investigate the safety and effectiveness of the AXIOS™ lumen-apposing Metal Stent used in the EUS-guided double-balloon-occluded gastrojejunostomy bypass (EPASS) for the management of symptoms associated with gastric outlet obstruction (GOO) secondary to malignant unresectable neoplasm.

Primary Endpoint is GOOSS 3 rate without MAE at 30 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable malignant duodenal obstruction confirmed by biopsy
* Eligible for endoscopic intervention
* GOOSS score of 0 or 1
* 18 years of age or older
* Willing and able to comply with the study procedures or legally authorized representative (LAR) must provide written informed consent form (ICF) to participate in the study

Exclusion Criteria:

* GOO symptoms are not expected to improve after the index procedure
* Life expectancy is about 3 months or less, which is not assumed applicable for surgical GJ
* Prior metallic stent placement for GOO
* Contraindicated to surgery and general anesthesia
* Neoplasm invading the target site of puncture in gastric and/or jejunum
* Abnormal coagulation INR > 1.5 and not correctable (per the discretion of the physician) or who require continuous complete anticoagulation
* Bleeding diathesis
* Altered anatomy of the upper gastrointestinal tract due to surgery of esophagus, stomach and duodenum that might preclude endoscopic drainage
* Presence of ileus caused by peritoneal carcinomatosis, or expected to present within 30 days post procedure
* Intervening gastric varices or vessels at the target site of stent insertion
* Ascites that may interfere the safety of the index procedure
* Biliary tract obstruction requiring treatment at the same day of the index procedure
* Allergic to any of the device materials
* Contraindications to use of electrosurgical devices
* Pregnancy, breastfeeding or intending to become pregnant during the study period
* Subject is currently participating, or plans to participate in, another investigational trial that may confound the results of this trial (unless written approval is received from the study sponsor)
* Vulnerable subject
* Subject has other reason not to be eligible for this study per investigators' discretion
* Guidewire doesn't cross the area of GOO
* EP-DB doesn't advance to the target site in jejunum
* The distance between the gastric wall and jejunal wall when visualized on ultrasound after saline is introduced into the space between the two inflated balloons of EP-DB is deemed about 2 cm or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
GOOSS 3 rate without MAE | 30 days post index-procedure
  GOOSS 3 rate without MAE

CONTACTS AND LOCATIONS:
Overall Officials: Takao Itoi, MD, Principal Investigator — Tokyo Medical University Hospital
Locations (6):
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
The anonymized data and study protocol for this clinical trial may be made available to other researchers in accordance with Boston Scientific Data Sharing Policy: (http://www.bostonscientific.com/en-US/data-sharing-requests.html)